CLINICAL TRIAL: NCT02221297
Title: Lowering Serum LDL-cholesterol With a Plant Stanol Ester Supplement Product
Brief Title: Lipid-lowering Effect of a Plant Stanol Ester Supplement Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Raisio Group (Industry)
Collaborators: Clinical Research Institute HUCH Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL2014_035
Record Dates: First submitted 2014-08-19; First posted 2014-08-20 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Hypercholesterolemia; Hyperlipidemias; Dyslipidemias
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias; Dyslipidemias | interventions — plant stanol ester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Supplement product with plant stanol ester (Experimental)
  Interventions: Dietary Supplement: Supplement product with plant stanol ester
- Placebo supplement product (Placebo Comparator)
  Interventions: Dietary Supplement: Supplement product with plant stanol ester

INTERVENTIONS:
Dietary Supplement: Supplement product with plant stanol ester — 2 grams plant stanols consumed with a meal daily for 3 to 4 weeks

SUMMARY:
Purpose of the study is to determine the effect of the investigational products as consumed with a meal on serum lipids, primarily on LDL cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* male and female over 18 years old
* serum LDL cholesterol > 3.0 mmol/L
* BMI < 35
* subjects must voluntarily sign the informed consent

Exclusion Criteria:

* subjects using lipid lowering medication (ezetimibe, bile acid sequestrant, statin therapy)
* subjects with any hepatic or renal disorder according to medical history
* subjects who have history of myocardial infarction or unstable angina pectoris within six months prior to screening
* subjects who have history of coronary artery bypass graft or percutaneous transluminal coronary angioplasty within six months prior to screening
* subjects who have history of temporal ischemic attack or stroke within six months prior to screening
* subjects who have a history of cancer or other malignant disease within the past five years
* subjects who are consuming more than 15 portions of alcohol / week
* subjects who are pregnant or lactating
* subjects using cholesterol-lowering foods or dietary supplements within 14 days before start of the intervention
* subjects with intolerance to any ingredient of the test product

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2014-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Proportional change in serum LDL cholesterol | 3 to 4 weeks
  Proportional change [end of intervention - start of intervention] in serum LDL-cholesterol between intervention and control groups in subjects fulfilling the inclusion criteria at the beginning of the study.

SECONDARY OUTCOMES:
Proportional change in total cholesterol | 3 to 4 weeks
  Proportional change [end of intervention - start of intervention] in serum total cholesterol between intervention and control groups in subjects fulfilling the inclusion criteria at the beginning of the study.
Proportional change in non-HDL-cholesterol | 3 to 4 weeks
  Proportional change [end of intervention - start of intervention] in serum non-HDL-cholesterol between intervention and control groups in subjects fulfilling the inclusion criteria at the beginning of the study.
Proportional change in serum triglycerides | 3 to 4 weeks
  Proportional change [end of intervention - start of intervention] in serum triglycerides between intervention and control groups in subjects fulfilling the inclusion criteria at the beginning of the study.
Proportional change in lipids in all study participants | 3 to 4 weeks
  Proportional change [end of intervention - start of intervention] in serum lipids in all study participants (ITT analysis)
Proportional change in lipids in subjects without metabolic derangements | 3 to 4 weeks
  Proportional change [end of intervention - start of intervention] in serum lipids in study participants without metabolic derangements (excluding those with type two diabetes and/or metabolic syndrome)